CLINICAL TRIAL: NCT00007631
Title: CSP #402 - VA Topical Tretinoin Chemoprevention Trial
Brief Title: Determine the Efficacy of Topical Tretinoin Cream for the Prevention of Nonmelanoma Skin Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Ortho Dermatologics (Industry)
Responsible Party: Weinstock, Martin - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 402
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Skin Neoplasms
Keywords: NMSC; nonmelanoma skin cancer; topical tretinoin cream
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Skin Neoplasms | interventions — Tretinoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Topical Tretinoin
  Interventions: Drug: Tretinoin 0.1% cream or placebo
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tretinoin 0.1% cream or placebo
  Arms: 1
Other: Placebo — Patients receive placebo for same amount of time
  Arms: 2

SUMMARY:
One-third of all malignancies in the United States (approximately one million cases diagnosed annually) are nonmelanoma skin cancer (NMSC). NMSC causes considerable morbidity, economic burden, facial deformity and at least 1,000 deaths annually. Prevention of these malignancies with a topical agent free of serious side effects would confer substantial public health benefit. Three hundred fifty thousand veterans were expected to develop NMSC in 1994. NMSC is one of the most common conditions requiring dermatologic care in the VA system. Topical tretinoin has been used extensively to treat photoaged skin. Retinoids administered orally in high doses appear to be effective in chemoprevention of nonmelanoma skin cancer but have unacceptable toxicity. In this study, 1131 patients with a recent history of squamous cell and/or basal cell carcinoma were enrolled at six participating centers over a four-year period and were randomly assigned to either 0.1% tretinoin cream or placebo. They were followed for a minimum of two years to determine if topical tretinoin is effective in reducing the risk of new occurrences.

DETAILED DESCRIPTION:
Primary Hypothesis: To determine the efficacy of topical tretinoin cream for the prevention of nonmelanoma skin cancer (NMSC) among high risk individuals (at least 2 NMSC?S in last 5 years).

Secondary Hypothesis: Secondary objectives are: (a) to determine the long-term effect of topical tretinoin on the prevalence of premalignant actinic keratoses, and (b) to distinguish subpopulations in which topical tretinoin is particularly effective or ineffective, compared to the overall study population.

Intervention: Apply Tretinoin 0.1% cream or placebo cream to face and ears twice a day.

Primary Outcomes: New NMSC lesions on the face and ears. Number of actinic keratoses on the face and ears.

Study Abstract: One-third of all malignancies in the United States (approximately one million cases diagnosed annually) are nonmelanoma skin cancer (NMSC). NMSC causes considerable morbidity, economic burden, facial deformity and at least 1,000 deaths annually. Prevention of these malignancies with a topical agent free of serious side effects would confer substantial public health benefit. Three hundred fifty thousand veterans were expected to develop NMSC in 1994. NMSC is one of the most common conditions requiring dermatologic care in the VA system.

Topical tretinoin has been used extensively to treat photoaged skin. Retinoids administered orally in high doses appear to be effective in chemoprevention of nonmelanoma skin cancer but have unacceptable toxicity. In this study, 1200 patients with a recent history of squamous cell and/or basal cell carcinoma will be enrolled at six participating centers over a four-year period and will be randomly assigned to either 0.1% tretinoin cream or placebo. They will be followed for a minimum of two years to determine if topical tretinoin is effective in reducing the risk of new occurrences.

Weinstock, M.A., Bingham, S.F., Cole, G.W., Eilers, D., Naylor, M.F., Kalivas, J., Taylor, J.R., Gladstone, H.B., Piacquadio, D.J., and DiGiovanna, J.J. Reliability of Counting Actinic Keratoses Before and After Brief Consensus Discussion. Arch Dermatol 137:1055-1058, 2001

ELIGIBILITY:
Inclusion Criteria:

High risk individuals (at least 2 NMSC?S in last 5 years).

Exclusion Criteria:

Exclusion criteria would include systemic retinoid treatment or systemic chemotherapy within the past six months; indices of very high mortality risk within 3 years (history of invasive noncutaneous malignancy within the past five years or metastatic cutaneous malignancy, or of other severe medical problems e.g. end-stage cardiac disease); known allergy or severe irritation reaction to tretinoin or the cream vehicle; special conditions predisposing to NMSC that may not be generally applicable (xeroderma pigmentosum, basal cell nevus syndrome, major organ transplant recipient, known arsenic exposure, PUVA photochemotherapy, mycosis fungoides, or prior or current radiation therapy involving the face, ears, or area of prior skin cancer), and likely inability to comply with the requirements of the trial as judged by the investigator. Incompetent patients and pregnant or nursing patients will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1131 (Actual)
Dates: Start 1998-03; Primary Completion 2004-11 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Long term effect of topical tretinoin on the prevalence of premalignant actinic keratoses | until the end of the study for a minimum of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin A. Weinstock, MD, Study Chair — VA Medical Center, Providence
Locations (7):
- United States (7):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - VA Medical Center, Long Beach, Long Beach, California
  - VA Medical Center, Miami, Miami, Florida
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Oklahoma City, Oklahoma City, Oklahoma
  - VA Medical Center, Providence, Providence, Rhode Island

REFERENCES:
- [Derived] Weinstock MA, Bingham SF, Lew RA, Hall R, Eilers D, Kirsner R, Naylor M, Kalivas J, Cole G, Marcolivio K, Collins J, Digiovanna JJ, Vertrees JE; Veterans Affairs Topical Tretinoin Chemoprevention (VATTC) Trial Group. Topical tretinoin therapy and all-cause mortality. Arch Dermatol. 2009 Jan;145(1):18-24. doi: 10.1001/archdermatol.2008.542. PMID 19153339
- [Derived] Dore DD, Lapane KL, Trivedi AN, Mor V, Weinstock MA. Association between statin use and risk for keratinocyte carcinoma in the veterans affairs topical tretinoin chemoprevention trial. Ann Intern Med. 2009 Jan 6;150(1):9-18. doi: 10.7326/0003-4819-150-1-200901060-00004. PMID 19124815